CLINICAL TRIAL: NCT05905679
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Study to Examine the Effects of a Probiotic on Aspects of Mental Wellness
Brief Title: Effects of a Probiotic on Aspects of Mental Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BIO-2306
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-06

CONDITIONS: Mental Health Wellness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Arm (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: Probiotics
- Placebo (Active Comparator)
  Interventions: Dietary Supplement: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Probiotics — 6 Billion CFU
  Arms: Probiotic Arm
Dietary Supplement: Dietary Supplement: Placebo — 0 CFU per day
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare the effect of a probiotic strain on mental wellbeing in moderately stressed, healthy, adults in the general population. The main question it aims to answer is

• what is the impact of probiotic consumption on overall mental wellbeing? Participants will consume one probiotic or placebo capsule per day, answer a set of questionnaire (at 3 time points) and wear a wearable device for the total duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at screening.
2. Score of ≥14 on the Perceived Stress Scale questionnaire.
3. Has access to a dedicated iPhone with iOS 12+ or an Android 8+ capable of downloading and running the study specific app.
4. Willing to maintain habitual diet and lifestyle, physical activity patterns, and body weight during the study period.
5. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
6. Has no plan to change nicotine habits during the study period.
7. Has no health conditions that would prevent her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
8. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Daily consumption of prebiotic, postbiotic, or probiotic supplements as well as foods/beverages fortified to contain live probiotics (e.g., kombucha) within 2 weeks of screening.
2. Clinically diagnosed neurologic or psychiatric disorders (e.g., bipolar disorder, clinical depression, post-partum depression) currently requiring medication, such as antipsychotics, anticonvulsants, and antiparkinsonian agents as well as medications for bipolar disorder.
3. Current use of prescription stimulant medications [e.g., amphetamines/dextroamphetamine (Adderall), methylphenidate (Ritalin, Concerta), methamphetamine (Desoxyn), dextroamphetamine (Dexedrine), lisdexamfetamine (Vyvanse)].
4. Current use of antibiotics.
5. Clinically diagnosed GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, Crohn's disease, celiac disease).
6. Use of cannabis, marijuana or cannabinoid products, including those that are consumed, orally inhaled, smoked, applied topically, etc. within 6 months of screening.
7. Contraindication or allergy/sensitivity to any components in the study product or allergens present in the facility used to manufacture or pack the study product (Appendix 7).
8. Elective hospitalizations planned (e.g., elective cosmetic procedures) during the study period.
9. Exposure to any non-registered drug product within 4 weeks of screening.
10. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
11. Recent history of (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
12. Has a condition the Clinical Investigator believes would interfere with the subject's ability to provide informed consent, comply with the study protocol, confound the interpretation of the study results, or put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change in Mental wellbeing | 4 weeks
  Improvement in mental wellbeing will be measured using the Oxford Happiness Questionnaire (OHQ).
  The Oxford Happiness Inventory was devised as a broad measure of personal happiness. The OHQ has a total of 29 items. Each item is scored on a Likert scale from 1 to 6 (1=strongly disagree; 2=moderately disagree; 3=slightly disagree; 4=slightly agree; 5=moderately agree; 6=strongly agree). Some items are phrased positively and others negatively. Such that negative items (1, 3, 12, 13, 16, 18, 21 and 29) should be scored in reverse (Hills & Argyle, 2002). The total score is then divided by 29. Interpretation of the final score is as follows: A final score between 1 to 2 is considered "not happy"; between 2 and 3 is "somewhat unhappy"; between 3 and 4 is considered "Neutral"; 4 is "somewhat or moderately happy"; between 4 and 5 is "rather happy"; between 5 and 6 is "very happy"; 6 is "too happy".

SECONDARY OUTCOMES:
Change in Stress scores | 4 weeks
  Change in stress scores will be measured using the short version of the Depression, Anxiety, Stress Scale (DASS-21). Each item is scored from 0 to 3, with a score of 0 indicating that the statement did not apply or never. A score of 3 indicates that the statement applied very much or almost always. In DASS-21, items 1, 6, 8, 11, 12, 14 and 18 relate to measurement of stress. Given that DASS-21 is the short version of DASS-42, the total item score is multiplied by 2. The final total scores range from 0 (no stress) to 42 (extremely stressed). Scores ranging between 0-14 (stress) are considered normal. Scores above 14 are considered positive for stress.
Change in anxiety scores | 4 weeks
  Change in anxiety scores will be measured using the short version of the Depression, Anxiety, Stress Scale (DASS-21). Each item is scored from 0 to 3, with a score of 0 indicating that the statement did not apply or never. A score of 3 indicates that the statement applied very much or almost always. In DASS-21, items 2, 4, 7, 9, 15, 19 and 20 relate to measurement of anxiety. Given that DASS-21 is the short version of DASS-42, the total item score is multiplied by 2. The final total scores range from 0 (no anxiety) to 42 (extremely anxious). Scores ranging between 0-14 (stress) are considered normal. Scores above 14 are considered positive for anxiety.
Change in Depression scores | 4weeks
  Change in depression scores will be measured using the short version of the Depression, Anxiety, Stress Scale (DASS-21). Each item is scored from 0 to 3, with a score of 0 indicating that the statement did not apply or never. A score of 3 indicates that the statement applied very much or almost always. In DASS-21, items 3, 5, 10, 13, 16, 17, and 21 relate to measurement of depression . Given that DASS-21 is the short version of DASS-42, the total item score is multiplied by 2. The final total scores range from 0 (no depression ) to 42 (extremely depressed). Scores ranging between 0-14 (stress) are considered normal. Scores above 14 are considered positive for depression .
Change in Stress Scores | 4 weeks
  In addition o the DASS, Subjects will complete the Perceived Stress Scale during screening for eligibility purposes and on Days 13 and 27 for outcome assessments. The Perceived Stress Scale is a retrospective 10-item questionnaire asking about feelings and thoughts "over the last month" . Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items.
  Eligible participants will be required to have a total score ≥14, indicating moderate (score 14-26) or high (27-40) perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn B Beckman,, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No